CLINICAL TRIAL: NCT00791778
Title: A Double-Blind, Randomized Phase II Study Evaluating the Efficacy and Safety of Sorafenib Compared to Placebo in Ovarian Epithelial Cancer or Primary Peritoneal Cancer Patients Who Have Achieved a Complete Clinical Response After Standard Platinum/Taxane Containing Chemotherapy
Brief Title: Comparison of Nexavar/Placebo as Maintenance Therapy for Patients With Advanced Ovarian or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12007; 2008-004429-41 (EudraCT Number)
Record Dates: First submitted 2008-11-14; First posted 2008-11-17 (Estimated); Results first posted 2012-11-30 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-06

CONDITIONS: Ovarian Neoplasms
Keywords: Peritoneal Neoplasma
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sorafenib (Nexavar, BAY43-9006) (Experimental): Participants received 2 sorafenib tablets (200 mg each) per oral twice daily (bid)
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)
- Placebo (Placebo Comparator): Participants received 2 matching placebo tablets per oral twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — Patients in Sorafenib arm will receive 2 Sorafenib tablets (200 mg each) twice a day and in continuous administration.
  Arms: Sorafenib (Nexavar, BAY43-9006)
Drug: Placebo — Patients in Placebo arm will receive 2 matching placebo tablets twice a day and in continuous administration.
  Arms: Placebo

SUMMARY:
Comparison of Nexavar with a placebo as maintenance therapy for patients with advanced Ovarian or primary Peritoneal cancers in complete remission following surgery and one regimen of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed International Federation of Gynecology and Obstetrics (FIGO) stage (67) III or IV ovarian epithelial cancer or primary peritoneal cancer at presentation. Patients must have achieved a clinical complete response (disappearance of all clinical and radiological evidence of tumor) after only one regimen (4-6 cycles) of platinum and taxane-based standard chemotherapy received after tumor debulkment.
* Normal serum CA125 (cancer-associated tumor marker) level within 7 days of first dose of sorafenib.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* All scans used to document complete response must be done within 30 days prior to randomization.
* Patients must be able to swallow and retain oral medication.

Exclusion Criteria:

* Patients with any residual cancer tissue after the completion of chemotherapy detectable by standard Computed tomography (CT) or magnetic resonance imaging (MRI).
* Prior local radiotherapy, neoadjuvant chemotherapy or intraperitoneal chemotherapy.
* Histologic subtypes of ovarian cancer other than epithelial (i.e. sarcoma, lymphoma, germ cell).
* Major surgery, open biopsy, or significant traumatic injury within 30 days prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2008-11; Primary Completion 2011-07 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (51):
- United States (4):
  - La Jolla, California
  - Jacksonville, Florida
  - Augusta, Georgia
  - Scarborough, Maine
- Belgium (5):
  - Bruxelles - Brussel
  - Edegem
  - La Louvière
  - Leuven
  - Wilrijk
- Canada (4):
  - Hamilton, Ontario
  - London, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Finland (2):
  - Jyväskylä
  - Kuopio
- France (5):
  - Angers
  - Caen
  - Lyon
  - Tours
  - Villejuif
- Berlin, State of Berlin, Germany
- Hong Kong, Hong Kong
- Italy (4):
  - Meldola, Forlì
  - Campobasso
  - Milan
  - Roma
- Japan (6):
  - Nagoya, Aichi-ken
  - Kashiwa, Chiba
  - Isehara, Kanagawa
  - Shimotsuke, Tochigi
  - Koto-ku, Tokyo
  - Minato-ku, Tokyo
- Netherlands (2):
  - Maastricht
  - The Hague
- Poland (6):
  - Bialystok
  - Gdynia
  - Krakow
  - Lublin
  - Poznan
  - Warsaw
- Singapore, Singapore
- South Korea (6):
  - Seoul, Seoul Teugbyeolsi
  - Daegu
  - Gyeonggi-do
  - Incheon
  - Seoul
  - Sŏwŏn
- Spain (4):
  - Sabadell, Barcelona
  - Lugo, Lugo
  - Madrid, Madrid
  - Seville, Sevilla

REFERENCES:
- [Result] Herzog TJ, Scambia G, Kim BG, Lhomme C, Markowska J, Ray-Coquard I, Sehouli J, Colombo N, Shan M, Petrenciuc O, Oza A. A randomized phase II trial of maintenance therapy with Sorafenib in front-line ovarian carcinoma. Gynecol Oncol. 2013 Jul;130(1):25-30. doi: 10.1016/j.ygyno.2013.04.011. Epub 2013 Apr 13. PMID 23591401
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Period: Double-blind Treatment
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Started | 123 | 123
Completed | 46 (includes: 42 subjects with progression, 4 subjects transferred to a continuation study) | 75 (includes: 75 subjects with progression)
Not Completed | 77 | 48
Not completed — Adverse Event | 49 | 9
Not completed — Physician Decision | 6 | 26
Not completed — Protocol Violation | 0 | 4
Not completed — Withdrawal by Subject | 20 | 9
Not completed — Non-compliant with study medication | 2 | 0
Period: Follow-up
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Started | 100 | 91
Completed | 95 (Includes 79 participants with study follow-up terminated by sponsor and 16 deaths) | 90 (Includes 78 participants with study follow-up terminated by sponsor and 12 deaths)
Not Completed | 5 | 1
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo | Total
Number analyzed (Participants) | 123 | 123 | 246
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.9 (10.4) | 54.4 (10.3) | 55.7 (10.4)
Age, Customized [Number; unit: Participants]
  < 65 years | 95 | 99 | 194
  ≥ 65 - < 75 years | 23 | 23 | 46
  ≥ 75 years | 5 | 1 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 123 | 246
  Male | 0 | 0 | 0
Performance status, Eastern Cooperative Oncology Group (ECOG) [Number; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status is a scale that measures how cancer affects the daily life of a patient on an ordinal scale from grade 0 (best) to grade 5 (worst).
  Participants
    0=Fully active without restriction | 89 | 92 | 181
    1=Restricted in physically strenuous activity | 32 | 30 | 62
    2=Ambulatory, capable of all selfcare | 1 | 0 | 1
    Missing | 1 | 1 | 2
Type of cancer [Number; unit: Participants] — Patients were to have either ovarian epithelial cancer or primary peritoneal cancer. Primary peritoneal carcinoma involves the extra-ovarian peritoneum significantly and the ovarian surface minimally or not at all.
  Participants
    Ovarian cancer | 115 | 114 | 229
    Peritoneal cancer | 8 | 9 | 17
Previous Intra-peritoneal (IP) chemotherapy [Number; unit: Participants] — The presence or absence of any IP chemotherapy before enrollment into the study.
  Participants
    Yes | 5 | 4 | 9
    No | 118 | 119 | 237
Surgical cytoreduction [Number; unit: Participants] — The degree of residual disease following initial diagnosis and surgical debulkment: optimal surgical cytoreduction (any/each lesion remaining after surgery ≤1 cm) or suboptimal surgical cytoreduction (any/each lesion remaining after surgery >1cm)
  Participants
    Optimal | 105 | 105 | 210
    Suboptimal | 10 | 10 | 20
    Missing | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS), Based on Radiological or Pathologic Assessment
Description: Time from randomization to the first documented disease progression by radiological or pathologic assessment or death due to any cause whichever occurred first. For patients who had not progressed or died at the time of analysis, PFS was censored at the date of their last evaluable tumor scan.
Time Frame: From randomization of the first patient until 32.5 months later, assessed every 8 weeks
Population: Full analysis set (FAS)=all randomized participants
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 123 | 123
Days | 386 [230 to 691] | 478 [337 to 567]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; Sample size based on the primary efficacy endpoint of PFS. Clinically meaningful improvement defined as 65% increase in median PFS. With one-sided alpha of 0.10, power of 90% and a randomization ratio of 1:1 between Sorafenib and Placebo, a total of 105 PFS events were required; Test type: Superiority or Other; p = 0.655, Log Rank; Two treatment groups compared using a log-rank test with one-sided alpha of 0.10 stratified by the same factors as randomization; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.72 to 1.63] — Sorafenib compared to Placebo

2. Secondary Outcome: Time to First Pathologic CA-125 (Cancer-associated Tumor Marker) Serum Level
Description: Time from randomization to the first documented increase of CA-125 above the upper limit of normal. Patients without pathologic CA-125 increase at the time of analysis were censored at their last date of evaluation of CA-125.
Time Frame: From randomization of the first patient until 32.5 months later, assessed every 8 weeks
Population: Per protocol set (PPS)=all randomized participants who had normal CA-125 serum level at baseline and at least one post-baseline CA-125 assessment
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 119 | 111
Days | 337 [197 to NA] — Can't be estimated due to censored data. | 617 [392 to NA] — Can't be estimated due to censored data.
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; Test type: Superiority or Other; p = 0.951, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.43, 95% CI 2-sided [0.93 to 2.20] — Sorafenib compared to Placebo

3. Secondary Outcome: Overall Survival (OS)
Description: The OS time was measured from the date of randomization until the date of death due to any cause. Patients who were alive at the time of analysis were censored at the date of the last contact (last time the patient was known to be alive).
Time Frame: From randomization of the first patient until 32.5 months later
Population: FAS=all randomized participants
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 123 | 123
Days | NA [NA to NA] — Can't be estimated due to censored data. | NA [NA to NA] — Can't be estimated due to censored data.
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; Test type: Superiority or Other; p = 0.84, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.49, 95% CI 2-sided [0.69 to 3.23] — Sorafenib compared to Placebo

4. Other Pre Specified Outcome: Functional Assessment of Cancer Therapy (FACT)/National Comprehensive Cancer Network (NCCN) Ovarian Symptom Index (FOSI) Total Score at Cycle 1/Baseline
Description: The FOSI is an 8-item index derived from the FACT-Ovarian Cancer (FACT-O) to measure symptom response to treatment for ovarian cancer. The FOSI total score ranges from 0 (severely symptomatic) to 32 (asymptomatic).
Time Frame: At Cycle 1 (4 weeks per Cycle)/baseline
Population: Patient-reported outcomes (PRO) analysis set=the FAS population with evaluable PRO assessments at baseline and at least one post-baseline assessment
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 104 | 115
Scores on a scale | 25.909 (3.174) | 25.658 (3.968)

5. Other Pre Specified Outcome: FOSI Total Score at Cycle 3
Description: as for outcome 4
Time Frame: At Cycle 3 (4 weeks per Cycle)
Population: PRO analysis set=the FAS population with evaluable PRO assessments at baseline and at Cycle 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 70 | 105
Scores on a scale | 25.871 (3.166) | 26.105 (3.414)

6. Other Pre Specified Outcome: Change From Baseline in FOSI Total Score at Cycle 3
Description: The FOSI is an 8-item index derived from the FACT-Ovarian Cancer (FACT-O) to measure symptom response to treatment for ovarian cancer. The change is calculated as score at Cycle 3 minus baseline score. The change in FOSI total score ranges from -32 (most deterioration from baseline) to 32 (most improvement from baseline).
Time Frame: Baseline and Cycle 3 (4 weeks per Cycle)
Population: PRO analysis set=the FAS population with evaluable PRO assessments at baseline and at Cycle 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 70 | 105
Scores on a scale | 0.086 (3.387) | 0.460 (3.128)

7. Other Pre Specified Outcome: FOSI Total Score at Cycle 5
Description: as for outcome 4
Time Frame: At Cycle 5 (4 weeks per Cycle)
Population: PRO analysis set=the FAS population with evaluable PRO assessments at baseline and at Cycle 5
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 57 | 93
Scores on a scale | 25.496 (3.830) | 26.634 (2.922)

8. Other Pre Specified Outcome: Change From Baseline in FOSI Total Score at Cycle 5
Description: The FOSI is an 8-item index derived from the FACT-Ovarian Cancer (FACT-O) to measure symptom response to treatment for ovarian cancer. The change is calculated as score at Cycle 5 minus baseline score. The change in FOSI total score ranges from -32 (most deterioration from baseline) to 32 (most improvement from baseline).
Time Frame: Baseline and Cycle 5 (4 weeks per Cycle)
Population: PRO analysis set=the FAS population with evaluable PRO assessments at baseline and at Cycle 5
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 57 | 93
Scores on a scale | -0.223 (3.530) | 0.659 (3.380)

9. Other Pre Specified Outcome: FOSI Total Score at End of Treatment
Description: as for outcome 4
Time Frame: At End of treatment (up to Cycle 33, 4 weeks per Cycle)
Population: PRO analysis set=the FAS population with evaluable PRO assessments at baseline and at end of treatment
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 76 | 76
Scores on a scale | 25.011 (3.832) | 24.528 (3.579)

10. Other Pre Specified Outcome: Change From Baseline in FOSI Total Score at End of Treatment
Description: The FOSI is an 8-item index derived from the FACT-Ovarian Cancer (FACT-O) to measure symptom response to treatment for ovarian cancer. The change is calculated as score at End of treatment minus baseline score. The change in FOSI total score ranges from -32 (most deterioration from baseline) to 32 (most improvement from baseline).
Time Frame: Baseline and End of treatment (up to Cycle 33, 4 weeks per Cycle)
Population: PRO analysis set=the FAS population with evaluable PRO assessments at baseline and at end of treatment
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 76 | 76
Scores on a scale | -0.733 (4.089) | -1.088 (4.067)

11. Other Pre Specified Outcome: EuroQol-5D (EQ-5D) Index Score at Cycle 1/Baseline
Description: The EQ-5D contains a descriptive system which measures 5 health dimensions: mobility, self-care, usual activity, pain/discomfort, and anxiety/depression. These five health dimensions are summarized into a single score, the EQ-5D index score which ranges from -0.594 (worst) to 1 (best) when the United Kingdom (UK) weights are applied.
Time Frame: At Cycle 1 (4 weeks per Cycle)/baseline
Population: PRO analysis set=the FAS population with evaluable PRO assessments at baseline and at least one post-baseline assessment
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 104 | 116
Scores on a scale | 0.804 (0.168) | 0.779 (0.218)

12. Other Pre Specified Outcome: EQ-5D Index Score at Cycle 3
Description: as for outcome 11
Time Frame: At Cycle 3 (4 weeks per Cycle)
Population: PRO analysis set=the FAS population with evaluable PRO assessments at baseline and at Cycle 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 72 | 110
Scores on a scale | 0.727 (0.219) | 0.767 (0.232)

13. Other Pre Specified Outcome: Change From Baseline in EQ-5D Index Score at Cycle 3
Description: The EQ-5D contains a descriptive system which measures 5 health dimensions: mobility, self-care, usual activity, pain/discomfort, and anxiety/depression. These five health dimensions are summarized into a single score, the EQ-5D index. The change is calculated as score at Cycle 3 minus baseline score. The change in EQ-5D index ranges from -1.594 (most deterioration from baseline) to 1.594 (most improvement from baseline).
Time Frame: Baseline and Cycle 3 (4 weeks per Cycle)
Population: PRO analysis set=the FAS population with evaluable PRO assessments at baseline and at Cycle 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 72 | 110
Scores on a scale | -0.068 (0.225) | -0.003 (0.201)

14. Other Pre Specified Outcome: EQ-5D Index Score at Cycle 5
Description: as for outcome 11
Time Frame: At Cycle 5 (4 weeks per Cycle)
Population: PRO analysis set=the FAS population with evaluable PRO assessments at baseline and at Cycle 5
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 60 | 95
Scores on a scale | 0.744 (0.217) | 0.813 (0.159)

15. Other Pre Specified Outcome: Change From Baseline in EQ-5D Index Score at Cycle 5
Description: The EQ-5D contains a descriptive system which measures 5 health dimensions: mobility, self-care, usual activity, pain/discomfort, and anxiety/depression. These five health dimensions are summarized into a single score, the EQ-5D index. The change is calculated as score at Cycle 5 minus baseline score. The change in EQ-5D index ranges from -1.594 (most deterioration from baseline) to 1.594 (most improvement from baseline).
Time Frame: Baseline and Cycle 5 (4 weeks per Cycle)
Population: PRO analysis set=the FAS population with evaluable PRO assessments at baseline and at Cycle 5
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 60 | 95
Scores on a scale | -0.045 (0.222) | 0.016 (0.180)

16. Other Pre Specified Outcome: EQ-5D Index Score at End of Treatment
Description: as for outcome 11
Time Frame: At End of treatment (up to Cycle 33, 4 weeks per Cycle)
Population: PRO analysis set=the FAS population with evaluable PRO assessments at baseline and at end of treatment
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 76 | 72
Scores on a scale | 0.731 (0.235) | 0.741 (0.250)

17. Other Pre Specified Outcome: Change From Baseline in EQ-5D Index Score at End of Treatment
Description: The EQ-5D contains a descriptive system which measures 5 health dimensions: mobility, self-care, usual activity, pain/discomfort, and anxiety/depression. These five health dimensions are summarized into a single score, the EQ-5D index. The change is calculated as score at End of treatment minus baseline score. The change in EQ-5D index ranges from -1.594 (most deterioration from baseline) to 1.594 (most improvement from baseline).
Time Frame: Baseline and End of treatment (up to Cycle 33, 4 weeks per Cycle)
Population: PRO analysis set=the FAS population with evaluable PRO assessments at baseline and at end of treatment
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 76 | 72
Scores on a scale | -0.064 (0.243) | -0.054 (0.274)

18. Other Pre Specified Outcome: EQ-5D Visual Analogue Scale (VAS) Score at Cycle 1/Baseline
Description: The EQ-5D also contains a VAS, which records the respondent's self-rated health status on a vertical graduated scale. The scale ranges from 0 (worst imaginable health state) to 100 (best imaginable health state).
Time Frame: At Cycle 1 (4 weeks per Cycle)/baseline
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 102 | 114
Scores on a scale | 75.235 (14.494) | 75.868 (16.725)

19. Other Pre Specified Outcome: EQ-5D VAS Score at Cycle 3
Description: as for outcome 18
Time Frame: At Cycle 3 (4 weeks per Cycle)
Population: PRO analysis set=the FAS population with evaluable PRO assessments at baseline and at Cycle 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 71 | 109
Scores on a scale | 73.042 (14.701) | 77.899 (16.503)

20. Other Pre Specified Outcome: Change From Baseline in EQ-5D VAS Score at Cycle 3
Description: The EQ-5D also contains a VAS, which records the respondent's self-rated health status on a vertical graduated scale. The change is calculated as score at Cycle 3 minus baseline score. The change in EQ-5D VAS ranges from -100 (most deterioration from baseline) to 100 (most improvement from baseline).
Time Frame: Baseline and Cycle 3 (4 weeks per Cycle)
Population: PRO analysis set=the FAS population with evaluable PRO assessments at baseline and at Cycle 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 71 | 109
Scores on a scale | -2.225 (15.594) | 2.688 (10.736)

21. Other Pre Specified Outcome: EQ-5D VAS Score at Cycle 5
Description: as for outcome 18
Time Frame: At Cycle 5 (4 weeks per Cycle)
Population: PRO analysis set=the FAS population with evaluable PRO assessments at baseline and at Cycle 5
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 57 | 94
Scores on a scale | 75.404 (14.177) | 79.915 (16.339)

22. Other Pre Specified Outcome: Change From Baseline in EQ-5D VAS Score at Cycle 5
Description: The EQ-5D also contains a VAS, which records the respondent's self-rated health status on a vertical graduated scale. The change is calculated as score at Cycle 5 minus baseline score. The change in EQ-5D VAS ranges from -100 (most deterioration from baseline) to 100 (most improvement from baseline).
Time Frame: Baseline and Cycle 5 (4 weeks per Cycle)
Population: PRO analysis set=the FAS population with evaluable PRO assessments at baseline and at Cycle 5
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 57 | 94
Scores on a scale | -0.947 (15.901) | 3.543 (14.151)

23. Other Pre Specified Outcome: EQ-5D VAS Score at End of Treatment
Description: as for outcome 18
Time Frame: At End of treatment (up to Cycle 33, 4 weeks per Cycle)
Population: PRO analysis set=the FAS population with evaluable PRO assessments at baseline and at end of treatment
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 75 | 69
Scores on a scale | 71.413 (16.686) | 76.246 (16.017)

24. Other Pre Specified Outcome: Change From Baseline in EQ-5D VAS Score at End of Treatment
Description: The EQ-5D also contains a VAS, which records the respondent's self-rated health status on a vertical graduated scale. The change is calculated as score at End of treatment minus baseline score. The change in EQ-5D VAS ranges from -100 (most deterioration from baseline) to 100 (most improvement from baseline).
Time Frame: Baseline and End of treatment (up to Cycle 33, 4 weeks per Cycle)
Population: PRO analysis set=the FAS population with evaluable PRO assessments at baseline and at end of treatment
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 75 | 69
Scores on a scale | -2.147 (18.054) | 0.348 (17.481)

ADVERSE EVENTS:
Time Frame: From the start of treatment up to 30 days after last study drug administration.
Description: Acronyms used: Gastrointestinal (GI), Genitourinary (GU), Not Otherwise Specified (NOS), Absolute Neutrophil Count (ANC), Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), Common Terminology Criteria for Adverse Events (CTCAE)
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Serious Adverse Events (participants affected / at risk) | 26/123 | 25/123
Other Adverse Events (participants affected / at risk) | 121/123 | 105/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (Nexavar, BAY43-9006) (N=123) | Placebo (N=123)
Neutrophils (Blood and lymphatic system disorders) | 0 | 1
Hemoglobin (Blood and lymphatic system disorders) | 1 | 0
Lymphatics - Other (Blood and lymphatic system disorders) | 1 | 0
SupraVentricular arrhythmia, Atrial fibrillation (Cardiac disorders) | 2 | 0
Hypertension (Cardiac disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Fistula, GI, Colon/Cecum/Appendix (Gastrointestinal disorders) | 1 | 0
Mucositis (functional/symptomatic), Esophagus (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 1
Obstruction, GI, Ileum (Gastrointestinal disorders) | 0 | 1
Obstruction, GI, Small bowel NOS (Gastrointestinal disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 1 | 0
Fever (General disorders) | 2 | 0
Pain, Back (General disorders) | 0 | 1
Pain, Chest/thorax NOS (General disorders) | 1 | 0
Pain, Abdomen NOS (General disorders) | 2 | 1
Pain, Head/headache (General disorders) | 1 | 0
Pain, Other (Specify) (General disorders) | 0 | 1
Pain, Kidney (General disorders) | 0 | 1
Syndromes - Other (General disorders) | 0 | 1
No Code In CTCAE (General disorders) | 0 | 6
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Liver dysfunction (Hepatobiliary disorders) | 1 | 0
Allergic reaction (Immune system disorders) | 1 | 0
Allergy - Other (Immune system disorders) | 1 | 0
Infection (Documented clinically), Urinary tract NOS (Infections and infestations) | 1 | 0
Infection with normal ANC, Urinary tract NOS (Infections and infestations) | 1 | 0
Intraop injury - Other (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Musculoskeletal and connective tissue disorders) | 1 | 4
Secondary Malignancy (possibly related to cancer treatment) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mood Alteration, Anxiety (Nervous system disorders) | 1 | 0
Neurology - Other (Nervous system disorders) | 2 | 0
Syncope (fainting) (Nervous system disorders) | 1 | 1
Fistula, GU, Vagina (Renal and urinary disorders) | 1 | 0
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 3 | 0
Wound complication, non-infectious (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatology - Other (Skin and subcutaneous tissue disorders) | 1 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3 | 1
Ulceration (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Thrombosis/embolism (vascular access) (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (Nexavar, BAY43-9006) (N=123) | Placebo (N=123)
Neutrophils (Blood and lymphatic system disorders) | 12 | 8
Platelets (Blood and lymphatic system disorders) | 9 | 0
Leukocytes (Blood and lymphatic system disorders) | 10 | 3
Edema: Limb (Blood and lymphatic system disorders) | 4 | 14
Hypertension (Cardiac disorders) | 45 | 8
Tinnitus (Ear and labyrinth disorders) | 7 | 1
Anorexia (Gastrointestinal disorders) | 20 | 5
Constipation (Gastrointestinal disorders) | 24 | 18
Diarrhea (Gastrointestinal disorders) | 48 | 22
Gastritis (Gastrointestinal disorders) | 7 | 6
Heartburn (Gastrointestinal disorders) | 6 | 9
Mucositis (functional/symptomatic), Oral cavity (Gastrointestinal disorders) | 25 | 7
Nausea (Gastrointestinal disorders) | 33 | 26
GI - Other (Gastrointestinal disorders) | 8 | 10
Vomiting (Gastrointestinal disorders) | 22 | 17
Fever (General disorders) | 11 | 10
Insomnia (General disorders) | 8 | 8
Fatigue (General disorders) | 38 | 28
Pain, Back (General disorders) | 10 | 16
Pain, Extremity - limb (General disorders) | 11 | 15
Pain, Abdomen NOS (General disorders) | 21 | 20
Pain, Head/headache (General disorders) | 29 | 19
Pain, Joint (General disorders) | 13 | 17
Pain, Muscle (General disorders) | 7 | 9
Pain, Other (Specify) (General disorders) | 7 | 11
Pain, Pain NOS (General disorders) | 10 | 5
Pain, Stomach (General disorders) | 7 | 8
Pain, Throat/pharynx/larynx (General disorders) | 7 | 2
Flu-like syndrome (General disorders) | 11 | 16
Allergic reaction (Immune system disorders) | 7 | 3
Infection (Documented clinically), Upper airway NOS (Infections and infestations) | 5 | 7
Infection - Other (Infections and infestations) | 7 | 3
Infection with unknown ANC, Upper airway NOS (Infections and infestations) | 4 | 7
ALT (Metabolism and nutrition disorders) | 13 | 6
AST (Metabolism and nutrition disorders) | 12 | 7
Hypokalemia (Metabolism and nutrition disorders) | 7 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 8 | 1
Metabolic/Lab - Other (Metabolism and nutrition disorders) | 9 | 4
Musculoskeletal - Other (Musculoskeletal and connective tissue disorders) | 10 | 9
Dizziness (Nervous system disorders) | 9 | 6
Neuropathy: sensory (Nervous system disorders) | 16 | 15
Cystitis (Renal and urinary disorders) | 3 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 13
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 9 | 11
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 6 | 8
Voice changes (Respiratory, thoracic and mediastinal disorders) | 13 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 14 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 13 | 15
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 81 | 17
Dermatology - Other (Skin and subcutaneous tissue disorders) | 22 | 11
Pruritus (Skin and subcutaneous tissue disorders) | 24 | 11
Rash/desquamation (Skin and subcutaneous tissue disorders) | 62 | 18
Flushing (Skin and subcutaneous tissue disorders) | 10 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 7 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less